CLINICAL TRIAL: NCT03380897
Title: Sleep Disturbances and Depression of the Mother Affect to the Pain During Balloon Catheter Induction of Labour
Brief Title: Sleep and Depression in Induction of Labour
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: University of Turku (Other)
Responsible Party: Principal Investigator, Kirsi Rinne, Senior Doctor, Turku University Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: T146/2017
Record Dates: First submitted 2017-05-30; First posted 2017-12-21 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Prolonged Pregnancy; Sleep Disturbance; Depression
Keywords: induction of labor; double balloon catheter; mechanical ripening
MeSH Terms: conditions — Pregnancy, Prolonged; Parasomnias; Depression | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Factorial assignment
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Outpatient group (Active Comparator): After insertion of induction catheter for labor, women of the outpatient group can go home and assess their pain with visual analogy scale at home. The intervention is to go home.
  Intervention for outpatient group was to go home.
  Interventions: Other: Intervention for outpatient group was to go home
- Inpatient group (Placebo Comparator): After insertion of induction catheter for labor, women of the inpatient group assess their pain with visual analogy scale in the ward. The intervention is to stay at ward.
  Intervention for inpatient group was to stay at ward.
  Interventions: Other: Intervention for inpatient group was to stay at ward

INTERVENTIONS:
Other: Intervention for outpatient group was to go home — Intervention for outpatient group was to go home and assess the the pain
  Other Names: Intervention was to assess the pain by visual analogy scale.
  Arms: Outpatient group
Other: Intervention for inpatient group was to stay at ward — Intervention for inpatient group was to stay at ward and assess the pain
  Other Names: Intervention was to assess the pain by visual analogy scale.
  Arms: Inpatient group

SUMMARY:
Randomised trial comparing double balloon catheter for induction of labor between inpatient and outpatient groups. The investigators assess how sleep disturbances and depression of the mother affect to the pain during balloon catheter induction of labour.

DETAILED DESCRIPTION:
Participants included to this randomised study are women with uncomplicated singleton pregnancy with ≥ 37- ≤ 41+5 weeks of gestation. Participants are randomised to two groups: one hundred are randomised to the inpatient and one hundred to the outpatient group.

The main outcome measure is the pain evaluated by VAS at one, five , nine and 13 hours after the placement of double balloon induction catheter. The investigators assess also the effect of the sleep disturbance and depression of the mother to the pain during balloon catheter induction of the labour.

The total hospital stay and induction to delivery interval time is measured. Also the mode of birth as well as maternal and neonatal morbidity and patient satisfaction are recorded.

ELIGIBILITY:
Inclusion Criteria:

* uncomplicated pregnancy
* singleton pregnancy
* pregnancy weeks ≥ 37 - ≤ 41+5
* the patient is living in1/2 hour away from hospital

Exclusion Criteria:

* patient has a disease that is effecting to the pregnancy e.g. pre-eclampsia, gestational hepatosis
* the patient has medical treatment of diabetes
* baby is not growing normally
* multiple pregnancy
* preterm rupture of membranes
* earlier caesarean section
* the patient is living more than 1/2 hour away from hospital

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 117 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
The pain measured by VAS | one to 14 days after induction of the labor
  The pain measured by VAS after double balloon catheter insertion.

SECONDARY OUTCOMES:
The affect of the sleep disturbances of the mother to the pain assessed by VAS | one to 14 days after induction of the labor
  The affect of the sleep disturbances to the pain assessed by VAS
The effect of depression of the mother to the pain assessed by VAS | one to 14 days after induction of the labor
  The effect of depression of the mother to the pain assessed by VAS
The total hospital stay in both groups | one to 14 days after induction of the labor
  The total hospital stay in both groups
The maternal and neonatal morbidity after balloon catheter induction | one to 14 days after induction of the labor
  The maternal and neonatal morbidity after balloon catheter induction

CONTACTS AND LOCATIONS:
Overall Officials: Kirsi M Rinne, PhD, Principal Investigator — Turku University Hospital; Päivi ML Polo, PhD, Study Director — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: No
Letter to patients

REFERENCES:
- [Result] Henry A, Madan A, Reid R, Tracy SK, Austin K, Welsh A, Challis D. Outpatient Foley catheter versus inpatient prostaglandin E2 gel for induction of labour: a randomised trial. BMC Pregnancy Childbirth. 2013 Jan 29;13:25. doi: 10.1186/1471-2393-13-25. PMID 23356673
- [Result] Sciscione AC, Muench M, Pollock M, Jenkins TM, Tildon-Burton J, Colmorgen GH. Transcervical Foley catheter for preinduction cervical ripening in an outpatient versus inpatient setting. Obstet Gynecol. 2001 Nov;98(5 Pt 1):751-6. doi: 10.1016/s0029-7844(01)01579-4. PMID 11704164
- [Result] Prager M, Eneroth-Grimfors E, Edlund M, Marions L. A randomised controlled trial of intravaginal dinoprostone, intravaginal misoprostol and transcervical balloon catheter for labour induction. BJOG. 2008 Oct;115(11):1443-50. doi: 10.1111/j.1471-0528.2008.01843.x. Epub 2008 Aug 19. PMID 18715244